CLINICAL TRIAL: NCT02998294
Title: Respiratory Volume Measure Using ExSpiron 1Xi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1-2016-0008
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: ICU(Intensive Care Unit) Patients; Mechanical Ventilation After Surgery
MeSH Terms: interventions — Ventilators, Mechanical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Respiratory monitoring group (Experimental)
  Interventions: Device: Respiratory Volume Monitor(RVM); Device: artificial respirator

INTERVENTIONS:
Device: Respiratory Volume Monitor(RVM) — The purpose of this study was to determine the accuracy of one-time respiratory volume measured by RVM compared to the one-time respiratory volume measured by mechanical ventilation in post-operative ICU patients.
  Other Names: ExSpiron™ 1Xi
Device: artificial respirator — The purpose of this study was to determine the accuracy of one-time respiratory volume measured by RVM compared to the one-time respiratory volume measured by mechanical ventilation in post-operative ICU patients.

SUMMARY:
The purpose of this study was to determine the accuracy of one-time respiratory volume measured by RVM(Respiratory Volume Monitor) compared to the one-time respiratory volume measured by mechanical ventilation in post-operative ICU patients.

DETAILED DESCRIPTION:
The purpose of this study was to determine the accuracy of one-time respiratory volume measured by RVM(Respiratory Volume Monitor) compared to the one-time respiratory volume measured by mechanical ventilation in post-operative ICU patients.

In addition, the investigators investigated the decrease in respiratory volume in opioid infusion after ventilator weaning in this patient, and to measure the one-time respiratory volume change by RVM during deep breathing induction using Inspirometry exercise.

ELIGIBILITY:
Inclusion Criteria:

* An adult patients ( ≥ age 19)
* patients who receive mechanical ventilation in the ICU of the Severance Hospital after surgery and plans to wean the mechanical ventilation within 3 days.

Exclusion Criteria:

* severe respiratory illness patients (pneumothorax, chest tube intubation status, severe restrictive respiratory disease, unilateral lung ventilation, lung transplantation status, chronic restrictive respiratory disease, hydrothorax, diaphragmatic movement disorder)
* If the candidate can not understand and carry out the experiment contents and process

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Respiratory volume measure using ExSpiron 1Xi | during 10-minute
  During mechanical ventilator, we obtained respiratory parameter from ventilator and also we collected same parameter via RVM.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided